CLINICAL TRIAL: NCT00036127
Title: Study of Alternate Formulation of Aripiprazole in Agitated Patients With Schizophrenic Disorders
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Purpose: Treatment
Other Study IDs: CN138-050
Record Dates: First submitted 2002-05-07; First posted 2002-05-09 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2007-09

CONDITIONS: Schizophrenia
Keywords: agitated schizophrenic patients
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

INTERVENTIONS:
Drug: aripiprazole

SUMMARY:
Study to learn if the alternate formulation is effective in agitated schizophrenic patients

ELIGIBILITY:
Inclusion Criteria:

* Agitated schizophrenic patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-04; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Local Institution, Anaheim, California
  - Local Institution, Cerritos, California
  - Local Institution, Chula Vista, California
  - Local Institution, Rosemead, California
  - Local Institution, San Diego, California
  - Local Institution, Atlanta, Georgia
  - Local Institution, Macon, Georgia
  - Local Instituton, Hoffman Estates, Illinois
  - Local Institution, Las Vegas, Nevada
  - Local Institution, Nashua, New Hampshire
  - Local Institution, New York, New York
  - Local Institution, Beachwood, Ohio
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Charleston, South Carolina
  - Local Institution, Houston, Texas
  - Local Institution, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Tran-Johnson TK, Sack DA, Marcus RN, Auby P, McQuade RD, Oren DA. Efficacy and safety of intramuscular aripiprazole in patients with acute agitation: a randomized, double-blind, placebo-controlled trial. J Clin Psychiatry. 2007 Jan;68(1):111-9. doi: 10.4088/jcp.v68n0115. PMID 17284138